CLINICAL TRIAL: NCT05558319
Title: GEM21menos65. A Phase III Trial for NDMM Patients Who Are Candidates for ASCT Comparing Extended VRD Plus Early Rescue Intervention vs Isatuximab-VRD vs Isatuximab-V-Iberdomide-D
Brief Title: NDMM Patients Candidates for ASCT Comparing Extended VRD Plus vs. Isa-VRD vs. Isa-V-Iberdomide
Acronym: GEM21menos65
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: PETHEMA Foundation (Other)
Collaborators: Bristol-Myers Squibb (Industry); Sanofi (Industry); Adknoma (Unknown); Start from scratch (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GEM21menos65
Record Dates: First submitted 2022-09-23; First posted 2022-09-28 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Newly Diagnosed Multiple Myeloma
MeSH Terms: interventions — Bortezomib; isatuximab; iberdomide; Lenalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control arm (A) (Active Comparator): INDUCTION: Isatuximab + VRD, 4 cycles. Isatuximab (IV) 10 mg/Kg, 1st cycle D: 1,8,15, 22. Cycles 2-4: D 1,15. Bortezomib (SC) 1.3 mg/m2, D:1, 4, 8, 11. Lenalidomide (PO) 25mg, D:1-21. Dexamethasone (PO) 40 mg, D: 1-4, 9-12.
  ASCT. The conditioning regimen is melphalan 200 mg/m2.
  CONSOLIDATION: Isatuximab + VRD, 2 cycles. Isatuximab (IV) 10 mg/Kg. D 1-15. Bortezomib (SC) 1.3 mg/m2, D:1, 4, 8, 11. Lenalidomide (PO) 25mg, D:1-21. Dexamethasone (PO) 40 mg, D: 1-4, 9-12.
  CONTINUOUS TREATMENT: Lenalidomide and monthly Isatuximab until progression, unacceptable toxicity, patient withdrawal, loss to follow up or death. During continuous treatment, dexamethasone 40 mg is used as a standardized premedication for Isatuximab.
  Interventions: Drug: Bortezomib; Drug: Isatuximab; Drug: Lenalidomide; Drug: Dexamethasone
- EXPERIMENTAL ARM (B): Extended VRD and Early Rescue Intervention (Experimental): INDUCTION: Includes two experimental lines:
  1. VRD extended to 18 cycles: Induction (VRDx6): Bortezomib (SC) 1.3 mg/m2, D: 1, 4, 8, and 11 (Q4W). Lenalidomide 25 mg (PO), D: 1-21 (Q4W). Dexamethasone 40 mg (PO) D 1 to 4 and 9 to 12 (Q4W). Isatuximab (IV) 10 mg/kg, D: 1, 8, 15, and 22 (Q4W) and D: 1-15 in subsequent cycles.
  2. Early detection of treatment failure and Early Rescue Intervention (ERI): Isatuximab-Iberdomide-Dexamethasone in continuous treatment. Isatuximab (IV) 10mg/kg Cycle 1: Days 1, 8, 15, and 22 (Q4W). Cycles 2 onwards: Days 1 and 15 (Q4W). Isatuximab will be infused monthly after 1 year treatment (Day 1 Q4W) including ASCT. Iberdomide (PO) 1,6 mg. D: 1-21 (Q4W). Dexamethasone (PO) 40 mg. D: 1, 8, 15, and 22 (Q4W).
  ASCT. The conditioning regimen is melphalan 200 mg/m2. CONSOLIDATION (VRDx2)- Extended VRD: VDx10, followed by lenalidomide plus dexamethasone maintenance.
  CONTINUOUS TREATMENT: Lenalidomide 15 mg, D: 1-21, and dexamethasone 20 mg, D: 1-4 (Q4W).
  Interventions: Drug: Bortezomib; Drug: Isatuximab; Drug: Iberdomide; Drug: Lenalidomide; Drug: Dexamethasone
- EXPLORATORY ARM (C) (Experimental): INDUCTION: Iberdomide plus Isatuximab, bortezomib and dexamethasone (four cycles). Isatuximab (IV) 10 mg/kg D 1, 8, 15, and 22 in the first Q4W; and days 1-15 in subsequent cycles. Iberdomide (PO) at 1.6 mg on days 1-21 of every 4-week cycle. Bortezomib (SC) at 1.3 mg/m2 on days 1, 4, 8, and 11 of every 4-week cycle. Dexamethasone 40 mg (PO) D 1-4, 9-12 (Q4W).
  ASCT. The conditioning regimen is melphalan 200 mg/m2.
  CONSOLIDATION: two cycles (Q4W) of Isatuximab, Iberdomide, Bortezomib and Dexamethasone, as in induction, starting approximately 2 months after hospital discharge or 3 months after transplantation. Isatuximab will be infused monthly since the start of continuous therapy (after the second cycle of consolidation).
  CONTINUOUS TREATMENT: Iberdomide and monthly Isatuximab until progression, unacceptable toxicity, patient withdrawal, loss to follow up or death. During continuous treatment, dexamethasone 40 mg is used as a standardized premedication for Isatuximab.
  Interventions: Drug: Bortezomib; Drug: Isatuximab; Drug: Iberdomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Bortezomib — Bortezomib
Drug: Isatuximab — Isatuximab
Drug: Iberdomide — Iberdomide
  Arms: EXPERIMENTAL ARM (B): Extended VRD and Early Rescue Intervention; EXPLORATORY ARM (C)
Drug: Lenalidomide — Lenalidomide
  Arms: Control arm (A); EXPERIMENTAL ARM (B): Extended VRD and Early Rescue Intervention
Drug: Dexamethasone — Dexamethasone

SUMMARY:
This is a Phase III open-label, 3-arm, parallel, randomized, controlled trial. The allocation ratio 1:1:1 and outcome assessment are blind to group allocation. Patients will be randomized from 3 arms. Patients will receive VRD extended + ASCT plus ERI or Isatuximab-VRD + ASCT or Isatuximab-VID + ASCT.

DETAILED DESCRIPTION:
Patients will receive induction treatment, which will consist: arm A (Isatuximab-VRD + ASCT) or arm B (VRD extended + ASCT plus ERI) or arm C (Isatuximab-VID + ASCT). After ASTC, patients will start consolidation which will be 2 cycles of similar treatment to induction.

Continuous treatment will follow after consolidation and patients will receive:

* arm A: Lenalidomide and monthly Isatuximab until progression, unacceptable toxicity, patient withdrawal, loss to follow up or death. During continuous treatment, dexamethasone 40 mg is used as a standardized premedication for Isatuximab.
* arm B: after 6 cycles of induction VRD, ASCT and two consolidation VRDs, treatment continues with 10 additional cycles of VRD. During the extension cycles, VRD changes the bortezomib and dexamethasone regimen. In these10 cycles, both bortezomib and dexamethasone will be administered, at the same doses as the previous ones, but on a weekly schedule, on days 1, 8, 15 and 22 of each cycle. The lenalidomide regimen remains unchanged.
* arm C: Iberdomide and monthly Isatuximab until progression, unacceptable toxicity, patient withdrawal, loss to follow up or death. During continuous treatment, dexamethasone 40 mg is used as a standardized premedication for Isatuximab.

The primary objective is to compare the efficacy of extended VRD + ASCT plus ERI (Arm B) vs. Isatuximab-VRD + ASCT (Arm A) in terms of proportion of patients who are MRD-negative by next generation flow cytometry (NGF) after 18 cycles + ASCT.

The primary endpoint, the MRD rate, takes as a reference the evaluation after the last extended VRD cycle, this is: 6 cycles for induction, 6 months for transplantation, 2 cycles for consolidation and 10 cycles until completing the 18 cycles of VRD, (in total about 24 months). For this reason,the primary endpoint in Arms A and C are established after a similar treatment time, which includes 4 cycles of induction, ASCT, 2 cycles of consolidation and 12 cycles of continuous treatment with Iberdomide plus Isatuximab (Dexamethasone to be determined).In patients of Arm B included in ERI, due to the great variability of the possible moments of incorporation in this therapeutic program, only rules are established for the moment and the realization or not of the transplant. The evaluation of the results will be carried out separately in the patients included, butalso in conjunction with the rest of the patients in Arm B to know the effect of the global strategy.

After the evaluation of the primary endpoint, continuous/maintenance treatment continues in Arms A, B and C, including patients in ARM B assigned to the ERI program. Obtaining conventional CR in either arm will require a BM analysis for MRD. In the case of stable response or improvement without RC, MRD controls have been pre-established. Due to the lack of data on tolerance and adherence to long-term treatment with Isatuximab and Iberdomide, changes in the therapeutic programs, for this reason, a complete revision of the therapeutic program has been predetermined at the moment in which the last patient included in the clinical trial reaches 36 months of treatment. At this point, taking into account the updated knowledge about continuous or maintenance treatments, the strategies for a second clinical trial or an extension of this clinical trial will be defined.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is, in the investigator's opinion, willing and able to comply with the protocol requirements.
2. Patient must be able to understand the study procedures.
3. Patient has given voluntary written informed consent before performance of any studyrelated procedure non part of normal medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to their future medical care.
4. Newly diagnosed multiple myeloma patient who requires start active treatment according to the 2014 IMWG criteria, namely clonal bone marrow plasma cells ≥10% or biopsy-proven bony or extramedullary plasmacytoma and any one or more of the following myeloma defining events: evidence of end organ damage that can be attributed to the underlying plasma cell proliferative disorder, specifically: Hypercalcaemia, Anaemia, Renal Insufficiency, or Bone lesions (one or more osteolytic lesions on skeletal radiography, CT, or PET-CT), and any one or more of the following biomarkers: clonal BMPC% ≥60%, i/u free light ratio ≥100 or > 1 focal lesions on MRI or PET/CT) [Lancet Oncol. 2014;15(12): e538-e548].
5. Patient must have a measurable secretory disease defined as either serum monoclonal protein of ≥ 0,5 g/dl or urine monoclonal (light chain) protein ≥ 200 mg/24 h. For patients whose disease is only measurable by serum FLC, the involved FLC should be ≥ 10mg/dL (100 mg/L), with an abnormal serum FLC ratio.
6. Patient must have an Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2.
7. Patient must be ≤ 65 years of age.
8. Patient must have adequate organ function, defined as follows:

   * Absolute neutrophil count (ANC) ≥1.0 X 109/L without G-CSF use in the prior 7 days
   * Hemoglobin ≥8.0 g/dL (prior red blood cell (RBC) transfusion or recombinant human erythropoietin use is permitted)
   * Platelets ≥ 75 x 109/L in participants in whom <50% of bone marrow nucleated cells are plasma cells and ≥ 50×109/L in participants in whom ≥50% of bone marrow nucleated cells are plasma cells (without transfusion support or thrombopoietin receptor agonist within 7 days before the laboratory test).
   * Calcium Corrected serum calcium ≤13.5 mg/dL (≤3.4 mmol/L); or free ionized calcium ≤6.5 mg/dL (≤1.6 mmol/L).
   * Total bilirubin ≤2 X ULN
   * ALT ≤2.5 X ULN
   * AST ≤2.5 X ULN
   * Renal: eGFRa: ≥40 mL/min/ 1.73 m2
   * Cardiac: LVEF (echo) ≥ 50%
9. Female patient: contraceptive use should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies. A female patient is eligible to participate if she is not pregnant or breastfeeding, and at least one of the following conditions applies:

   * Is not a woman of childbearing potential (WOCBP), i.e., fertile, following menarche and until becoming post-menopausal unless permanently sterile. Permanent sterilization methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy OR
   * Is a WOCBP and

     * She understands the potential teratogenic risk to the unborn child
     * She understands the need for effective contraception as stated in the protocol, without interruption, 28 days before starting study treatment, throughout the entire duration of study treatment, during dose interruptions and for at least 28 days after the last dose of study treatment.
     * She understands and agrees to inform the Investigator if a change or stop of method of contraception is needed.
     * She must be capable of complying with effective contraceptive measures.
     * She is informed and understands the potential consequences of pregnancy and the need to notify her study doctor immediately if there is a risk of pregnancy.
     * She understands the need to commence study treatment as soon as it is dispensed following a negative pregnancy test.
     * She understands and accepts the need to undergo pregnancy testing based on the frequency outlined in this plan and in the Informed Consent.
     * She acknowledges she understands the hazards iberdomide or lenalidomide can cause to an unborn fetus and the necessary precautions associated with the use of study drugs.

   The Investigator must ensure that a WOCBP: i) Complies with the conditions of the pregnancy prevention plan, including confirmation that she has an adequate level of understanding. ii) Acknowledges the aforementioned requirements.

   A WOCBP must have a negative highly sensitive serum pregnancy test (as required by local regulations) within 72 hours before the first dose of study drug.

   Nonchildbearing potential is defined as follows (by other than medical reasons):
   * Has not achieved menarche at some point.
   * Has undergone a hysterectomy or bilateral oophorectomy.
   * Has been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (ie, has had menses at any time in the preceding 24 consecutive months).
10. Male patient: contraceptive use should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

    Male patient is eligible to participate if he agrees to the following from the time of first dose of study until 6 months after the last dose of iberdomide or lenalidomide to allow for clearance of any altered sperm:
    * Understand the potential teratogenic risk if engaged in sexual activity with a pregnant female or a WOCBP.
    * Understand the need for the use of a condom even if he has had a vasectomy, if engaged in sexual activity with a pregnant female or a FCBP
    * Understand the potential teratogenic risk, so the subject should not donate semen or sperm.. Understand that the effects on fertility are currently unknown, therefore all family planning options and/or alternatives should be thoroughly discussed with the study doctor prior to receiving iberdomide.
11. All prior treatment-related toxicities (defined by National Cancer Institute- Common Toxicity Criteria for Adverse Events (NCI-CTCAE), version 5.0 must be ≤ Grade 1 at the time of enrolment except for alopecia.

Exclusion Criteria:

1. Patient has a diagnosis of primary amyloidosis, monoclonal gammopathy of undetermined significance (MGUS), smoldering multiple myeloma (SMM), plasma cell leukemia or active POEMS syndrome at the time of screening.
2. Patient has had clinical evidence of central nervous system (CNS) or pulmonary leukostasis, disseminated intravascular coagulation, or CNS multiple myeloma.
3. Prior history of malignancies, other than multiple myeloma (except for basal or squamous cell carcinoma of the skin, carcinoma in situ of the cervix or the breast), unless the patient has been free of the disease for ≥ 5 years.
4. Any serious medical condition that places the subject at an unacceptable risk if he or she participates in this study; subjects with conditions requiring chronic steroid or immunosuppressive treatment, such as rheumatoid arthritis, multiple sclerosis and/or lupus, that likely need additional steroid or immunosuppressive treatments in addition to the study treatment.
5. Pregnant or breastfeeding females.
6. Men and women of reproductive potential who are not using effective contraceptive methods (double barrier method, intrauterine device, oral contraception).
7. Patient is simultaneously enrolled in other interventional clinical trial.
8. Patient has used an investigational drug within 28 days or five half-lives, whichever is longer, preceding the first dose of study drug.
9. Patient must not have received prior radiotherapy (except localized palliative radiotherapy for pain, palliation or fracture) within 2 weeks of start of study therapy. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis.
10. Major surgery (except kyphoplasty) ≤ 4 weeks prior to initiating protocol therapy.
11. Patient has peripheral neuropathy or neuropathic pain grade 1 with pain or ≥2, as defined by the National Cancer Institute Terminology Criteria for Adverse Events (NCI CTCAE) Version 5.0.
12. Patient evidence of cardiovascular risk including any of the following:

    * Myocardial infarction within 6 months before randomization, or an unstable or uncontrolled disease/condition related to or affecting cardiac function (eg, unstable angina, congestive heart failure, New York Heart Association Class III-IV).
    * Uncontrolled cardiac arrhythmia.
    * Screening 12-lead ECG showing a baseline interval QTcF> 470 msec (exception: subjects with pacemaker).
    * Patients with uncontrolled hypertension.
13. Patients who have current unstable liver or biliary disease defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, persistent jaundice, or cirrhosis. Note: Stable chronic liver disease (including Gilbert's syndrome or asymptomatic gallstones) or hepatobiliary involvement of malignancy is acceptable if otherwise meets entry criteria.
14. Presence of active renal condition (infection, requirement for dialysis or any other condition that could affect patient's safety). Participants with isolated proteinuria resulting from MM are eligible, provided they fulfil inclusion criteria.
15. Evidence of active mucosal or internal bleeding.
16. Any serious medical condition or psychiatric illness that would interfere in understanding of the informed consent form.
17. Uncontrolled endocrine diseases (i.e. diabetes mellitus, hypothyroidism or hyperthyroidism) (i.e. requiring relevant changes in medication within the last month, or hospital admission within the last 3 months).
18. Patient with acute diffuse infiltrative pulmonary disease and/or pericardial disease.
19. Patient with severe chronic obstructive pulmonary disease (COPD) or asthma with forced expiratory volume in the first minute (FEV1) less than 50%.
20. History of interstitial lung disease or ongoing interstitial lung disease.
21. Subject has gastrointestinal disease that may significantly alter the absorption of iberdomide and/or other oral study treatment.
22. Patient has an active infection requiring systemic antibiotic, antiviral, or antifungal treatment at the time of starting treatment.
23. Patient has known HIV infection.
24. Patient has positive hepatitis B surface antigen (HBsAg), or hepatitis B core antibody (HBcAb) at screening or within 3 months prior to first dose of study treatment.
25. Patient has positive hepatitis C antibody test result or positive hepatitis C RNA test result at screening or within 3 months prior to first dose of study treatment. Note: Participants with positive Hepatitis C antibody due to prior resolved disease can be enrolled, only if a confirmatory negative Hepatitis C RNA test is obtained. Note: Hepatitis RNA testing is optional and participants with negative Hepatitis C antibody test are not required.
26. Patient require concurrent administration of a strong inhibitor or inducer of cytochrome P450 (CYP3A4/5) (including within 14 days of initiating study treatment).
27. Patient has a known immediate or delayed hypersensitivity reaction or idiosyncratic reactions to iberdomide or drugs chemically related to iberdomide.
28. Patient has a known immediate or delayed hypersensitivity reaction or idiosyncratic reactions to isatuximab or drugs chemically related to isatuximab, hypersensitivity reactions, or idiosyncratic reactions to other molecular antibodies.
29. Patient has a known immediate or delayed hypersensitivity reaction or idiosyncratic reactions to lenalidomide or dexamethasone or drugs chemically related to lenalidomide or dexamethasone.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Efficacy in terms of patients who are MRD-negative by NGF | 24 months
  Percentage of patients who are MRD-negative by next generation flow cytometry (NGF) after 18 cycles + ASCT comparing the efficacy of extended VRD + ASCT plus ERI & (Arm B) vs. IsatuximabVRD + ASCT (Arm A).

SECONDARY OUTCOMES:
Frequency of adverse events (AEs) | Throughout the study. Approximately 78 months.
  Number of patients who presented AEs in each arm to perform safety analysis. NOTE: Due to the experimental nature of the Arm C combination Isatuximab-Iberdomide-Bortezomib-Dex, a safety analysis will be performed with the first 5 patients included in each arm as per section, a second one when 25 patients in each arm have completed 3 cycles of therapy, and subsequent ones might be required if considered by the Primary-Investigator, Co-Primary-Investigator, Co-coordinators and Co-Investigator.
Progression-Free Survival (PFS) | Throughout the study. Approximately 78 months
  Time from the start of treatment until the earliest date of documented disease progression or death due to any cause.

OTHER OUTCOMES:
Overall Response Rate (ORR) | Throughout the study. Approximately 78 months
  Percentage of participants with a confirmed partial response (PR) or better (PR, VGPR, CR, sCR).
Complete Response Rate (CRR) | Throughout the study. Approximately 78 months
  The percentage of participants with a confirmed complete response (CR) or better (stringent complete response (CR, sCR)).
Time to Response (TTR) | Throughout the study. Approximately 78 months
  Time from the start of treatment and the first documented evidence of response (PR or better) among participants who achieve confirmed PR or better.
Duration of Response (DoR) | Throughout the study. Approximately 78 months
  Time from first documented evidence of PR or better until progressive disease (PD) or death due to PD among participants who achieved PR or better.
Overall Survival (OS) | Throughout the study. Approximately 78 months
  Time from the start of treatment until the date of death due to any cause

CONTACTS AND LOCATIONS:
Overall Officials: Juan José Lahuerta Palacios, Dr, Study Chair — Hospital Universitario 12 de Octubre; Joan Bladé, Dr, Study Chair — Hospital Clinic of Barcelona; Mª Victoria Mateos, Dr, Study Chair — Hospital Clínico Universitario de Salamanca; Enrique M Ocio, Dr, Study Chair — Hospital Universitario Marqués de Valdecilla; Jesús San Miguel, Dr, Study Chair — Clínica Universitaria de Navarra
Locations (68):
- Spain (68):
  - Hospital Principe de Asturias, Alcalá de Henares, Madrid
  - Hospital Universitario Quirón Salud Madrid, Pozuelo de Alarcón, Madrid
  - Clinica Universidad Navarra (CUN), Pamplona, Navarre
  - Hospital General Universitario de Albacete, Albacete
  - Hospital Germans Trias i Pujol (ICO BADALONA), Badalona
  - Hospital Clinic i Provincial de Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitari Vall d´Hebron, Barcelona
  - ICO L´Hospitalet, Barcelona
  - Hospital Universitario de Cruces, Bilbao
  - Hospital Universitario de Burgos, Burgos
  - Complejo Hospitalario de Cáceres, Cáceres
  - Hospital Universitario de Cabueñes, Gijón
  - Hospital Universitari Dr. Josep Trueta (ICO Girona), Girona
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital Universitario de Guadalajara, Guadalajara
  - H.Universitario de Jerez de la Frontera, Jerez de la Frontera
  - Complejo Asistencial Universitario de León, León
  - Hospital Arnau de Vilanova (Lleida), Lleida
  - Hospital San Pedro, Logroño
  - Complejo Hospitalario Lucus Augusti, Lugo
  - Fundación Jiménez Díaz-Ute, Madrid
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital HLA Universitario Moncloa, Madrid
  - Hospital Universitario 12 de octubre, Madrid
  - Hospital Universitario Clínico San Carlos, Madrid
  - Hospital Universitario de Fuenlabrada, Madrid
  - Hospital Universitario de la Princesa, Madrid
  - Hospital Universitario Fundación Alcorcón, Madrid
  - Hospital Universitario HM Sanchinarro, Madrid
  - Hospital Universitario Infanta Leonor, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario La Zarzuela, Madrid
  - Hospital Universitario Puerta del Hierro, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Costa del Sol, Málaga
  - Hospital Regional de Málaga, Málaga
  - Hospital U Niversitario Virgen de La Victoria, Málaga
  - Hospital Universitario Rey Juan Carlos, Móstoles
  - H. Morales Meseguer, Murcia
  - H. Un. Virgen de la Arrixaca, Murcia
  - Hospital General Universitario Santa Lucía, Murcia
  - Complejo Hospitalario Universitario de Ourense, Ourense
  - Hospital Universitario Central de Asturias, Oviedo
  - Hospital Son Llatzer, Palma de Mallorca
  - Hospital Universitari Son Espases, Palma de Mallorca
  - Complejo Hospitalario de Navarra, Pamplona
  - Complejo Hospitalario de Pontevedra, Pontevedra
  - Hospital Clinico Universitario Salamanca, Salamanca
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna
  - Hospital Universitario de Donostia, San Sebastián
  - Hospital Universitario Infanta Sofía, San Sebastián de los Reyes
  - Complejo Hospitalario Universitario Nuestra Señora de la Candelaria, Santa Cruz de Tenerife
  - H. Universitario Marqués de Valdecilla, Santander
  - Complejo Hospitalario Santiago (CHUS), Santiago de Compostela
  - Hospital General de Segovia, Segovia
  - Complejo Hospitalario Regional Virgen Del Rocío, Seville
  - H. Universitario de Valme, Seville
  - Hospital Universitario Reina Sofía, Seville
  - Hospital Universitari de Tarragona Joan XXIII, Tarragona
  - Hospital Universitari Mutua Terrassa, Terrassa
  - Complejo Hospitalario de Toledo (Virgen de la Salud), Toledo
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital Universitari i Politecnic la Fe, Valencia
  - Hospital Universitario Dr. Peset Aleixandre, Valencia
  - H. U. Txagorritxu, Vitoria-Gasteiz
  - Hospital Clinico Universitario Lozano Blesa, Zaragoza
  - Hospital Universitario Miguel Servet, Zaragoza

REFERENCES:
- [Background] Durie BGM, Hoering A, Abidi MH, Rajkumar SV, Epstein J, Kahanic SP, Thakuri M, Reu F, Reynolds CM, Sexton R, Orlowski RZ, Barlogie B, Dispenzieri A. Bortezomib with lenalidomide and dexamethasone versus lenalidomide and dexamethasone alone in patients with newly diagnosed myeloma without intent for immediate autologous stem-cell transplant (SWOG S0777): a randomised, open-label, phase 3 trial. Lancet. 2017 Feb 4;389(10068):519-527. doi: 10.1016/S0140-6736(16)31594-X. Epub 2016 Dec 23. PMID 28017406
- [Background] Attal M, Lauwers-Cances V, Hulin C, Leleu X, Caillot D, Escoffre M, Arnulf B, Macro M, Belhadj K, Garderet L, Roussel M, Payen C, Mathiot C, Fermand JP, Meuleman N, Rollet S, Maglio ME, Zeytoonjian AA, Weller EA, Munshi N, Anderson KC, Richardson PG, Facon T, Avet-Loiseau H, Harousseau JL, Moreau P; IFM 2009 Study. Lenalidomide, Bortezomib, and Dexamethasone with Transplantation for Myeloma. N Engl J Med. 2017 Apr 6;376(14):1311-1320. doi: 10.1056/NEJMoa1611750. PMID 28379796
- [Background] Rosinol L, Oriol A, Rios R, Sureda A, Blanchard MJ, Hernandez MT, Martinez-Martinez R, Moraleda JM, Jarque I, Bargay J, Gironella M, de Arriba F, Palomera L, Gonzalez-Montes Y, Marti JM, Krsnik I, Arguinano JM, Gonzalez ME, Gonzalez AP, Casado LF, Lopez-Anglada L, Paiva B, Mateos MV, San Miguel JF, Lahuerta JJ, Blade J. Bortezomib, lenalidomide, and dexamethasone as induction therapy prior to autologous transplant in multiple myeloma. Blood. 2019 Oct 17;134(16):1337-1345. doi: 10.1182/blood.2019000241. PMID 31484647
- [Background] Rosinol L, Oriol A, Teruel AI, Hernandez D, Lopez-Jimenez J, de la Rubia J, Granell M, Besalduch J, Palomera L, Gonzalez Y, Etxebeste MA, Diaz-Mediavilla J, Hernandez MT, de Arriba F, Gutierrez NC, Martin-Ramos ML, Cibeira MT, Mateos MV, Martinez J, Alegre A, Lahuerta JJ, San Miguel J, Blade J; Programa para el Estudio y la Terapeutica de las Hemopatias Malignas/Grupo Espanol de Mieloma (PETHEMA/GEM) group. Superiority of bortezomib, thalidomide, and dexamethasone (VTD) as induction pretransplantation therapy in multiple myeloma: a randomized phase 3 PETHEMA/GEM study. Blood. 2012 Aug 23;120(8):1589-96. doi: 10.1182/blood-2012-02-408922. Epub 2012 Jul 12. PMID 22791289
- [Background] Rosinol L, Hebraud B, Oriol A, Colin AL, Rios Tamayo R, Hulin C, Blanchard MJ, Caillot D, Sureda A, Hernandez MT, Arnulf B, Mateos MV, Macro M, San-Miguel J, Belhadj K, Lahuerta JJ, Garelik MB, Blade J, Moreau P. Integrated analysis of randomized controlled trials evaluating bortezomib + lenalidomide + dexamethasone or bortezomib + thalidomide + dexamethasone induction in transplant-eligible newly diagnosed multiple myeloma. Front Oncol. 2023 Nov 2;13:1197340. doi: 10.3389/fonc.2023.1197340. eCollection 2023. PMID 38023148
- [Background] Lin P, Owens R, Tricot G, Wilson CS. Flow cytometric immunophenotypic analysis of 306 cases of multiple myeloma. Am J Clin Pathol. 2004 Apr;121(4):482-8. doi: 10.1309/74R4-TB90-BUWH-27JX. PMID 15080299
- [Background] van de Donk NW, Janmaat ML, Mutis T, Lammerts van Bueren JJ, Ahmadi T, Sasser AK, Lokhorst HM, Parren PW. Monoclonal antibodies targeting CD38 in hematological malignancies and beyond. Immunol Rev. 2016 Mar;270(1):95-112. doi: 10.1111/imr.12389. PMID 26864107
- [Background] Attal M, Richardson PG, Rajkumar SV, San-Miguel J, Beksac M, Spicka I, Leleu X, Schjesvold F, Moreau P, Dimopoulos MA, Huang JS, Minarik J, Cavo M, Prince HM, Mace S, Corzo KP, Campana F, Le-Guennec S, Dubin F, Anderson KC; ICARIA-MM study group. Isatuximab plus pomalidomide and low-dose dexamethasone versus pomalidomide and low-dose dexamethasone in patients with relapsed and refractory multiple myeloma (ICARIA-MM): a randomised, multicentre, open-label, phase 3 study. Lancet. 2019 Dec 7;394(10214):2096-2107. doi: 10.1016/S0140-6736(19)32556-5. Epub 2019 Nov 14. PMID 31735560
- [Background] Leypoldt LB, Besemer B, Asemissen AM, Hanel M, Blau IW, Gorner M, Ko YD, Reinhardt HC, Staib P, Mann C, Lutz R, Munder M, Graeven U, Peceny R, Salwender H, Jauch A, Zago M, Benner A, Tichy D, Bokemeyer C, Goldschmidt H, Weisel KC. Isatuximab, carfilzomib, lenalidomide, and dexamethasone (Isa-KRd) in front-line treatment of high-risk multiple myeloma: interim analysis of the GMMG-CONCEPT trial. Leukemia. 2022 Mar;36(3):885-888. doi: 10.1038/s41375-021-01431-x. Epub 2021 Nov 3. No abstract available. PMID 34732857
- [Background] Dimopoulos MA, Oriol A, Nahi H, San-Miguel J, Bahlis NJ, Usmani SZ, Rabin N, Orlowski RZ, Komarnicki M, Suzuki K, Plesner T, Yoon SS, Ben Yehuda D, Richardson PG, Goldschmidt H, Reece D, Lisby S, Khokhar NZ, O'Rourke L, Chiu C, Qin X, Guckert M, Ahmadi T, Moreau P; POLLUX Investigators. Daratumumab, Lenalidomide, and Dexamethasone for Multiple Myeloma. N Engl J Med. 2016 Oct 6;375(14):1319-1331. doi: 10.1056/NEJMoa1607751. PMID 27705267
- [Background] Lonial S, Dimopoulos M, Palumbo A, White D, Grosicki S, Spicka I, Walter-Croneck A, Moreau P, Mateos MV, Magen H, Belch A, Reece D, Beksac M, Spencer A, Oakervee H, Orlowski RZ, Taniwaki M, Rollig C, Einsele H, Wu KL, Singhal A, San-Miguel J, Matsumoto M, Katz J, Bleickardt E, Poulart V, Anderson KC, Richardson P; ELOQUENT-2 Investigators. Elotuzumab Therapy for Relapsed or Refractory Multiple Myeloma. N Engl J Med. 2015 Aug 13;373(7):621-31. doi: 10.1056/NEJMoa1505654. Epub 2015 Jun 2. PMID 26035255
- [Background] Moreau P, Masszi T, Grzasko N, Bahlis NJ, Hansson M, Pour L, Sandhu I, Ganly P, Baker BW, Jackson SR, Stoppa AM, Simpson DR, Gimsing P, Palumbo A, Garderet L, Cavo M, Kumar S, Touzeau C, Buadi FK, Laubach JP, Berg DT, Lin J, Di Bacco A, Hui AM, van de Velde H, Richardson PG; TOURMALINE-MM1 Study Group. Oral Ixazomib, Lenalidomide, and Dexamethasone for Multiple Myeloma. N Engl J Med. 2016 Apr 28;374(17):1621-34. doi: 10.1056/NEJMoa1516282. PMID 27119237
- [Background] Palumbo A, Chanan-Khan A, Weisel K, Nooka AK, Masszi T, Beksac M, Spicka I, Hungria V, Munder M, Mateos MV, Mark TM, Qi M, Schecter J, Amin H, Qin X, Deraedt W, Ahmadi T, Spencer A, Sonneveld P; CASTOR Investigators. Daratumumab, Bortezomib, and Dexamethasone for Multiple Myeloma. N Engl J Med. 2016 Aug 25;375(8):754-66. doi: 10.1056/NEJMoa1606038. PMID 27557302
- [Background] Stewart AK, Rajkumar SV, Dimopoulos MA, Masszi T, Spicka I, Oriol A, Hajek R, Rosinol L, Siegel DS, Mihaylov GG, Goranova-Marinova V, Rajnics P, Suvorov A, Niesvizky R, Jakubowiak AJ, San-Miguel JF, Ludwig H, Wang M, Maisnar V, Minarik J, Bensinger WI, Mateos MV, Ben-Yehuda D, Kukreti V, Zojwalla N, Tonda ME, Yang X, Xing B, Moreau P, Palumbo A; ASPIRE Investigators. Carfilzomib, lenalidomide, and dexamethasone for relapsed multiple myeloma. N Engl J Med. 2015 Jan 8;372(2):142-52. doi: 10.1056/NEJMoa1411321. Epub 2014 Dec 6. PMID 25482145
- [Background] Nooka AK, Kaufman JL, Muppidi S, Langston A, Heffner LT, Gleason C, Casbourne D, Saxe D, Boise LH, Lonial S. Consolidation and maintenance therapy with lenalidomide, bortezomib and dexamethasone (RVD) in high-risk myeloma patients. Leukemia. 2014 Mar;28(3):690-3. doi: 10.1038/leu.2013.335. Epub 2013 Nov 13. PMID 24220275
- [Background] Ahn JS, Jung SH, Yang DH, Bae SY, Kim YK, Kim HJ, Lee JJ. Patterns of relapse or progression after bortezomib-based salvage therapy in patients with relapsed/refractory multiple myeloma. Clin Lymphoma Myeloma Leuk. 2014 Oct;14(5):389-94. doi: 10.1016/j.clml.2014.02.004. Epub 2014 Feb 18. PMID 24630919
- [Background] Alegre A, Granda A, Martinez-Chamorro C, Diaz-Mediavilla J, Martinez R, Garcia-Larana J, Lahuerta JJ, Sureda A, Blade J, de la Rubia J, Fernandez-Ranada JM, San Miguel J; Spanish Registry of Transplants in Multiple Myelomas; Spanish Group of Hemopoietic Transplant (GETH); PETHEMA. Different patterns of relapse after autologous peripheral blood stem cell transplantation in multiple myeloma: clinical results of 280 cases from the Spanish Registry. Haematologica. 2002 Jun;87(6):609-14. PMID 12031917
- [Background] Fernandez de Larrea C, Jimenez R, Rosinol L, Gine E, Tovar N, Cibeira MT, Fernandez-Aviles F, Martinez C, Rovira M, Blade J. Pattern of relapse and progression after autologous SCT as upfront treatment for multiple myeloma. Bone Marrow Transplant. 2014 Feb;49(2):223-7. doi: 10.1038/bmt.2013.150. Epub 2013 Sep 30. PMID 24076551
- [Background] Zamarin D, Giralt S, Landau H, Lendvai N, Lesokhin A, Chung D, Koehne G, Chimento D, Devlin SM, Riedel E, Bhutani M, Babu D, Hassoun H. Patterns of relapse and progression in multiple myeloma patients after auto-SCT: implications for patients' monitoring after transplantation. Bone Marrow Transplant. 2013 Mar;48(3):419-24. doi: 10.1038/bmt.2012.151. Epub 2012 Aug 13. PMID 22890289
- [Background] Durie BG, Harousseau JL, Miguel JS, Blade J, Barlogie B, Anderson K, Gertz M, Dimopoulos M, Westin J, Sonneveld P, Ludwig H, Gahrton G, Beksac M, Crowley J, Belch A, Boccadaro M, Cavo M, Turesson I, Joshua D, Vesole D, Kyle R, Alexanian R, Tricot G, Attal M, Merlini G, Powles R, Richardson P, Shimizu K, Tosi P, Morgan G, Rajkumar SV; International Myeloma Working Group. International uniform response criteria for multiple myeloma. Leukemia. 2006 Sep;20(9):1467-73. doi: 10.1038/sj.leu.2404284. Epub 2006 Jul 20. PMID 16855634
- [Background] Kumar S, Paiva B, Anderson KC, Durie B, Landgren O, Moreau P, Munshi N, Lonial S, Blade J, Mateos MV, Dimopoulos M, Kastritis E, Boccadoro M, Orlowski R, Goldschmidt H, Spencer A, Hou J, Chng WJ, Usmani SZ, Zamagni E, Shimizu K, Jagannath S, Johnsen HE, Terpos E, Reiman A, Kyle RA, Sonneveld P, Richardson PG, McCarthy P, Ludwig H, Chen W, Cavo M, Harousseau JL, Lentzsch S, Hillengass J, Palumbo A, Orfao A, Rajkumar SV, Miguel JS, Avet-Loiseau H. International Myeloma Working Group consensus criteria for response and minimal residual disease assessment in multiple myeloma. Lancet Oncol. 2016 Aug;17(8):e328-e346. doi: 10.1016/S1470-2045(16)30206-6. PMID 27511158
- [Background] Blade J, Samson D, Reece D, Apperley J, Bjorkstrand B, Gahrton G, Gertz M, Giralt S, Jagannath S, Vesole D. Criteria for evaluating disease response and progression in patients with multiple myeloma treated by high-dose therapy and haemopoietic stem cell transplantation. Myeloma Subcommittee of the EBMT. European Group for Blood and Marrow Transplant. Br J Haematol. 1998 Sep;102(5):1115-23. doi: 10.1046/j.1365-2141.1998.00930.x. No abstract available. PMID 9753033
- [Background] Rajkumar SV, Buadi F. Multiple myeloma: new staging systems for diagnosis, prognosis and response evaluation. Best Pract Res Clin Haematol. 2007 Dec;20(4):665-80. doi: 10.1016/j.beha.2007.10.002. PMID 18070712
- [Background] Rajkumar SV, Harousseau JL, Durie B, Anderson KC, Dimopoulos M, Kyle R, Blade J, Richardson P, Orlowski R, Siegel D, Jagannath S, Facon T, Avet-Loiseau H, Lonial S, Palumbo A, Zonder J, Ludwig H, Vesole D, Sezer O, Munshi NC, San Miguel J; International Myeloma Workshop Consensus Panel 1. Consensus recommendations for the uniform reporting of clinical trials: report of the International Myeloma Workshop Consensus Panel 1. Blood. 2011 May 5;117(18):4691-5. doi: 10.1182/blood-2010-10-299487. Epub 2011 Feb 3. PMID 21292775
- [Background] Lahuerta JJ, Paiva B, Vidriales MB, Cordon L, Cedena MT, Puig N, Martinez-Lopez J, Rosinol L, Gutierrez NC, Martin-Ramos ML, Oriol A, Teruel AI, Echeveste MA, de Paz R, de Arriba F, Hernandez MT, Palomera L, Martinez R, Martin A, Alegre A, De la Rubia J, Orfao A, Mateos MV, Blade J, San-Miguel JF; GEM (Grupo Espanol de Mieloma)/PETHEMA (Programa para el Estudio de la Terapeutica en Hemopatias Malignas) Cooperative Study Group. Depth of Response in Multiple Myeloma: A Pooled Analysis of Three PETHEMA/GEM Clinical Trials. J Clin Oncol. 2017 Sep 1;35(25):2900-2910. doi: 10.1200/JCO.2016.69.2517. Epub 2017 May 12. PMID 28498784
- [Background] Ferrero S, Ladetto M, Drandi D, Cavallo F, Genuardi E, Urbano M, Caltagirone S, Grasso M, Rossini F, Guglielmelli T, Cangialosi C, Liberati AM, Callea V, Carovita T, Crippa C, De Rosa L, Pisani F, Falcone AP, Pregno P, Oliva S, Terragna C, Musto P, Passera R, Boccadoro M, Palumbo A. Long-term results of the GIMEMA VEL-03-096 trial in MM patients receiving VTD consolidation after ASCT: MRD kinetics' impact on survival. Leukemia. 2015 Mar;29(3):689-95. doi: 10.1038/leu.2014.219. Epub 2014 Jul 16. PMID 25027515
- [Background] Paiva B, Chandia M VM. No Title. In: Additional prognostic value of multiparameter flow cytometry minimal residual disease monitoring over complete response across the clinical course of multiple myeloma patients. 2014. p. 256.
- [Background] Landgren O, Lu SX, Hultcrantz M. MRD Testing in Multiple Myeloma: The Main Future Driver for Modern Tailored Treatment. Semin Hematol. 2018 Jan;55(1):44-50. doi: 10.1053/j.seminhematol.2018.03.001. Epub 2018 Mar 5. PMID 29759154
- [Background] Anderson KC, Auclair D, Kelloff GJ, Sigman CC, Avet-Loiseau H, Farrell AT, Gormley NJ, Kumar SK, Landgren O, Munshi NC, Cavo M, Davies FE, Di Bacco A, Dickey JS, Gutman SI, Higley HR, Hussein MA, Jessup JM, Kirsch IR, Little RF, Loberg RD, Lohr JG, Mukundan L, Omel JL, Pugh TJ, Reaman GH, Robbins MD, Sasser AK, Valente N, Zamagni E. The Role of Minimal Residual Disease Testing in Myeloma Treatment Selection and Drug Development: Current Value and Future Applications. Clin Cancer Res. 2017 Aug 1;23(15):3980-3993. doi: 10.1158/1078-0432.CCR-16-2895. Epub 2017 Apr 20. PMID 28428191
- [Background] Matyskiela ME, Zhang W, Man HW, Muller G, Khambatta G, Baculi F, Hickman M, LeBrun L, Pagarigan B, Carmel G, Lu CC, Lu G, Riley M, Satoh Y, Schafer P, Daniel TO, Carmichael J, Cathers BE, Chamberlain PP. A Cereblon Modulator (CC-220) with Improved Degradation of Ikaros and Aiolos. J Med Chem. 2018 Jan 25;61(2):535-542. doi: 10.1021/acs.jmedchem.6b01921. Epub 2017 Apr 20. PMID 28425720
- [Background] Bjorklund CC, Kang J, Amatangelo M, Polonskaia A, Katz M, Chiu H, Couto S, Wang M, Ren Y, Ortiz M, Towfic F, Flynt JE, Pierceall W, Thakurta A. Iberdomide (CC-220) is a potent cereblon E3 ligase modulator with antitumor and immunostimulatory activities in lenalidomide- and pomalidomide-resistant multiple myeloma cells with dysregulated CRBN. Leukemia. 2020 Apr;34(4):1197-1201. doi: 10.1038/s41375-019-0620-8. Epub 2019 Nov 12. No abstract available. PMID 31719682
- [Background] Amatangelo M, Bjorklund CC, Kang J, Polonskaia A, Viswanatha S, Thakurta A. Iberdomide (CC-220) Has Synergistic Anti-Tumor and Immunostimulatory Activity Against Multiple Myeloma in Combination with Both Bortezomib and Dexamethasone, or in Combination with Daratumumab in Vitro. Blood [Internet]. 2018 Nov 29;132(Supplement 1):1935. Available from: https://doi.org/10.1182/blood-2018-99-113383
- [Background] Sagar Lonial, Paul G. Richardson, Rakesh Popat, Edward Stadtmauer, Jeremy Larsen, Albert Oriol, Stefan Knop, Sundar Jagannath, Gordon Cook, Ashraf Z. Badros, Paula Rodríguez Otero, David S. Siegel, Tuong Vi Nguyen, Antonia Di Micco, Alpesh Amin, Min Chen, NWCJ van de D. No Title. In: IBERDOMIDE (IBER) IN COMBINATION WITH DEXAMETHASONE (DEX) AND DARATUMUMAB (DARA), BORTEZOMIB (BORT), OR CARFILZOMIB (CFZ) IN PATIENTS (PTS) WITH RELAPSED/REFRACTORY MULTIPLE MYELOMA (RRMM). 2021.
- [Background] Amatangelo M, Bjorklund C, Kang J, Mukhopadhyay A, Jiménez Nuñez MD, Wong L, et al. Preclinical and Translational Support for Clinical Development of Iberdomide in Combination with Proteasome Inhibitors: Mechanism of Synergy in Clinical Trial CC-220-MM-001. Blood [Internet]. 2020 Nov 5;136(Supplement 1):8-9. Available from: https://doi.org/10.1182/blood-2020-137710
- [Background] Amatangelo M, Bjorklund C, Ma P, Wollerman K, Pierceall W, Lonial S, et al. Preclinical and Translational Data Support Development of Iberdomide in Combination with CD38- and SLAMF7-Directed Monoclonal Antibodies: Evidence for Rational Combinations. Blood [Internet]. 2020 Nov 5;136(Supplement 1):9-10. Available from: https://doi.org/10.1182/blood-2020-137667
- [Background] van de Donk NWCJ, Popat R, Larsen J, Minnema MC, Jagannath S, Oriol A, et al. First Results of Iberdomide (IBER; CC-220) in Combination with Dexamethasone (DEX) and Daratumumab (DARA) or Bortezomib (BORT) in Patients with Relapsed/Refractory Multiple Myeloma (RRMM). Blood [Internet]. 2020 Nov 5;136(Supplement 1):16-7. Available from: https://doi.org/10.1182/blood-2020-137743